CLINICAL TRIAL: NCT04404517
Title: Correlation of Serum Adalimumab Levels at an Administration of 40 mg Weekly vs 80 mg Every Two Weeks
Acronym: IntnsificADA
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Principal Investigator, María Dolores Martín Arranz, PhD, Director, Hospital Universitario La Paz
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IntnsificADA
Record Dates: First submitted 2019-09-16; First posted 2020-05-27 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Inflammatory Bowel Diseases
Keywords: AntiTNF; Inflammatory Bowel Diseases; Adalimumab; Therapeutic drug monitoring
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Adalimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 40mg1w (Active Comparator): Adalimumab at an administration of 40 mg weekly for 6 weeks, followed by Adalimumab at an administration of 80 mg every two weeks
  Interventions: Drug: Adalimumab
- 80mg2w (Active Comparator): Adalimumab at an administration of 80 mg every two weeks
  Interventions: Drug: Adalimumab

INTERVENTIONS:
Drug: Adalimumab — Monoclonal antibody used in IBD treatment

SUMMARY:
RCT to evaluate possible pharmacokinetic differences between the two current regimes of intensified adalimumab administration.

DETAILED DESCRIPTION:
IBD patients in need of intensified adalimumab treatment will be randomized to receive 40mg sc weekly or 80mg sc every two weeks, and after 6 weeks of treatment each of the groups will be allocated to the other dosing regime. Adalimumab blood levels and other features such as specific drug antibodies and disease activity parameters will be compared between both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18y
* Intensified adalimumab regime at least 4 weeks prior to enrollment.
* Immunosuppressants are allowed if a stable dose for > 12w is maintained.
* Corticosteroids are allowed if they were initiated prior to enrollment and a stable dose is maintained.

Exclusion Criteria:

* Patients unable to understand study protocol, study procedures or not capacitated to give informed consent.
* Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
Adalimumab trough level | 12 weeks
  Drug levels will be measured during 12 weeks of treatment

SECONDARY OUTCOMES:
Antibodies to Adalimumab (ADA) | 12 weeks
  Antibodies to Adalimumab will be tested for 12 weeks of treatment
Clinical response for Ulcerative Colitis | 12 weeks
  Simple Clinical Colitis Activity Index (SCCAI) (for UC) refers to disease symptoms during the previous week. It is composed of six domains. After recording, the clinician-based SCCAI is able to categorize two types of patients: patients with inactive disease (SCCAI<5) and patients with active disease (SCCAI≥5).
Clinical response for Ulcerative colitis | 12 weeks
  Truelove Index (for UC), is composed of 6 variables. Clinical remission was defined as 1 or 2 stools per day without blood, absence of fever or tachycardia, a normal hemoglobin or "returning towards normal," a normal ESR or "returning towards normal," and gaining weight.
Clinical response for Crohn´s Disease | 12 weeks
  Harvey-Bradshaw Index (for CD) considers five parameters. For each parameter a specific score is assigned. A score below 5 is considered as clinical remission. A reduction of 3 points is considered as relevant to define clinical response.
Fecal calprotectin | 12 weeks
  Fecal calprotectin levels will be tested during the study
Blood acute phase reactants | 12 weeks
  Blood acute phase reactants will be tested during the study
QOL | 12 weeks
  Quality of life will be analysed using the Inflammatory Bowel Disease Questionnaire
Treatment Satisfaction | 12 weeks
  Treatment Satisfaction Questionnaire for Medication (TSQM)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Dolores Martin Arranz, PhD, Study Director — Hospital Universitario La Paz. IdiPaz. Universidad Autónoma de Madrid.
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrd, Spain

IPD SHARING:
Plan to Share IPD: No